CLINICAL TRIAL: NCT06978972
Title: Cognitive Stimulation Therapy for Residents With Dementia in Long-Term Facilities: A Quasi-Experimental Study
Brief Title: Cognitive Stimulation Therapy for Residents With Dementia in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Kentucky University (Other)
Collaborators: Ridgewood Health Campus (Unknown)
Responsible Party: Principal Investigator, Abigail Genevieve Halsey, Doctor of Occupational Therapy Student, Northern Kentucky University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#: 2562
Record Dates: First submitted 2025-05-02; First posted 2025-05-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dementia in Nursing Home
Keywords: Skilled nursing facilities; occupational engagement; cognitive functioning; Cognitive stimulation therapy; dementia; Group intervention; long-term care; geriatrics
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive stimulation therapy group (Experimental): The CST group will participate in a screening measure where they will perform the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) to assess for cognitive impairment. The participants will then participate in the Montreal Cognitive Assessment (MoCA) and the Observational Measurement of Engagement (OME) prior to and after the 7-week CST program. The group will receive CST, which is an evidence-based, cognitively stimulating therapeutic group intervention, two times per week for 7 weeks for 45 minutes. The general structure of each session will follow the CST Manual called "Making a Difference 1" and each participant will participate in an introduction, theme song, current affairs activity, the main activity (theme-based activities), and closure each session.
  Interventions: Other: Cognitive Stimulation Therapy

INTERVENTIONS:
Other: Cognitive Stimulation Therapy — CST is an evidence-based, cognitively stimulating therapeutic group intervention for individuals with mild-to-moderate dementia. Individuals participate in CST 2 times per week for 7 weeks. The CST sessions are administered by a variety of professionals who become certified through the St. Louis School of Medicine. The general structure of each session will follow the CST Manual called "Making a Difference 1". Each session will be based on a theme and will include an introduction, theme song, current affairs activity, the main activity (physical games, sounds, food, being creative, word and number games, team quizzes, orientation, current affairs, ect.), suggested activities for home, and closure. These sessions are highly structured and will follow the introduction, theme song, current affairs activity, the main activity, suggested activities for home, and closure organization strictly. The participants will spend 45 minutes in each session.

SUMMARY:
The goal of this experimental study was to evaluate whether cognitive stimulation therapy (CST) improved cognitive functioning and engagement levels in individuals with mild-to-moderate dementia residing in long-term care facilities. The study aimed to: 1) investigate the preliminary effect of CST on cognition and engagement in individuals with mild-to-moderate dementia, and 2) assess the feasibility of implementing CST in LTC facilities in the Cincinnati metropolitan area.

The main question the study answered was: Does CST improve cognitive functioning and increase engagement levels in individuals with mild-to-moderate dementia living in long-term care facilities?

Researchers conducted CST (structured, themed, grouped sessions with activites related to their childhood, sounds, word and number games, current affairs, being creative, word association, physical games, quizzes, and orientation) sessions to see if there was a significant increase in cognition and engagement after the 7 weeks of activites.

Participants received CST for 45 to 60 minutes twice weekly for 7 weeks, led by two doctor of occupational therapy students under the supervision of a licensed occupational therapist in the state of Indiana. Participants completed assessments before and after the 7-weeks to measure changes in cognitive function and engagement, along with participating in a screening assessment before the start of the study.

DETAILED DESCRIPTION:
This study was a quasi-experimental one group pretest-posttest designed to evaluate the significance of a 7-week CST program among residents of a long-term care facility with mild to moderate dementia. The primary aim was to investigate the preliminary effect of CST on cognition and engagement in individuals with mild-to-moderate dementia.

The study was conducted at Ridgewood Health Campus and aimed to enroll approximately 10 participants over an estimated period of 1 to 2 months. Recruitment was completed with one research team member meeting site staff, where she presented the study and prepared them to identify eligible individuals based on the inclusion criteria. Site staff then provided a list of potential participants and gave access to relevant medical records, which the research team reviewed before reaching out to potential participants and/or their legal representatives via email, phone, or in person.

Interested participants and their Powers of Attorney (POAs) received an informational handout explaining study expectations. If the POA expressed interest in participation, an electronic version of the informed consent form was provided and reviewed. Research team members were available to address questions via phone, email, Zoom, or in person. The signed consent forms were returned electronically or physically, and a copy was retained by the participant and/or their POA.

As 10 participants enrolled, they first completed a one-week screening period, followed by one week of pre-testing. The CST intervention was administered twice weekly for 45 minutes over 7 weeks, followed by a one-week post-intervention assessment period.

To ensure fidelity of the CST intervention, the Principal Investigator (PI) and Co-Investigators (Co-PIs) completed formal training through the North American Cognitive Stimulation Therapy Training Institute through Saint Louis University, School of Medicine. The CST practice manual was also followed strictly. The research team then collaborated closely with on-site staff to address concerns related to participant safety, treatment environment, or study procedures. In the event of an adverse event, the research team planned to follow all HIPAA and facility protocols and planned to report the incident to the PI.

Given the vulnerability of the participant population, the research team prioritized ethical considerations. All study materials, including the participant handout and consent forms, were written in plain language and at an appropriate reading level. Power of Attorneys were given adequate time and support to make informed decisions. Additionally, on-site staff (nursing staff and aides) who were familiar with the participants were present during sessions to help meet their individual needs and advocate on their behalf. Additionally, because occupational therapy students co-facilitated the CST sessions, a licensed occupational therapist was present for all sessions to ensure participant safety and to ensure proper implementation of the intervention.

Participation was entirely voluntary, and participants could withdraw from the study at any time without penalty or loss of benefits. Participants were able to decline individual sessions or activities without consequence. During evaluations, participants were able to skip any question they did not wish to answer. Data from assessments were included in the analysis only if at least 75% of items were completed per participant. If a participant attended greater than or equal to 50% of the scheduled sessions (7 out of 14 sessions), their data was retained for analysis. Data from participants who attended fewer than 7 sessions were planned to be included from analysis, and this was addressed in the final report.

CST has not been associated with harmful side effects in previous studies, suggesting minimal risk to participants. Nonetheless, the possibility of emotional discomfort or other adverse events remained. Psychological effects were monitored, and any incident was planned to be addressed promptly following institutional and facility procedures. A potential risk includes unintentional disclosure of identifiable information, although safeguards have been implemented to mitigate this.

Data collection was managed using an encrypted password-protected flash drive with encryption and a password-protected file folder. Participant names were linked to unique ID codes necessary for tracking consent and study progress. Only coded identifiers were used in outcome data collection. Names were recorded solely on consent forms and a separate secure document linking names to ID codes, which will be stored for six years in accordance with data retention policies. After this period, all physical and electronic data will be securely destroyed.

Access to data was and will continue to be restricted to the PI and four Collaborative Institutional Training Initiative program (CITI) certified research members. Electronic documents were stored on two secure, encrypted, and password-protected flash drives. All team members' laptops are password-protected and use two-factor authentication. Devices have been and will continue to be stored securely when not in use, and team members adhere to strict data security practices when in public settings. Physical copies of data are stored in a password-protected file folder and stored with the faculty advisor.

All study procedures comply with Northern Kentucky University's institutional ethical guidelines. All protocol changes were submitted to the Institutional Review Board (IRB) before the start of the intervention and were approved. Data management followed validated protocols with comprehensive quality control measures to ensure the integrity and confidentiality of all collected data.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Adults aged 18 years or older who reside in a long-term care facility
* Adequate English proficiency, vision, hearing, and speech to participate in groups
* English proficiency
* participation in recreational or social activities for at least 45 minutes per week
* diagnosis of mild-to-moderate dementia based on Diagnostic and Statistical Manual of Mental Disorders (5th ed.; DSM-5) criteria, confirmed by medical records, or a mid-range score (18-55) on the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)

Exclusion Criteria:

* Prior CST treatment
* non-English speaking
* Communication barriers (aphasia)
* Diagnosis of severe dementia
* History of a learning disability or traumatic brain injury
* Participation in a concurrent clinical trial
* Receiving hospice care
* ADAS-Cog score in the no-impairment range (0-17) or high range (56-70).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | From/after the completion of enrollment (middle to end of June 2025) to after the completion of the 7-week CST sessions (week of August 18th).
  The MoCA assesses multiple areas of cognition such as attention, orientation, delayed recall, working memory, executive functioning, visuospatial, and language. The MoCA will take approximately 10 minutes to administer. MoCA scores range from 0 to 30, with higher scores indicating better cognitive functioning. Scores between 10 and 25 typically reflect mild to moderate cognitive impairment, and a score within this range is required for study inclusion. Therefore, only participants scoring between 10 and 25 at baseline will be enrolled, and we will assess whether their cognitive functioning improves from this initial range over the seven weeks.
The Observational Measurement of Engagement - OME Modified | From/after the completion of enrollment (middle to end of June 2025) to after the completion of the 7-week CST sessions (week of August 18th).
  The OME is a measurement tool used for individuals with dementia to document direct observations regarding their level of engagement during an activity. The OME assesses an individual's response to the stimuli during an activity by taking note of their attention and attitude using a rating scale. The OME also assesses the individual's cognitive and fine motor difficulty during the task, as well as, the duration and frequency of interactions in the task to determine overall engagement. The OME will take between 3 and 15 minutes to administer. Three minutes if the participant is disengaged with the stimulus and 15 minutes if the participant is engaged the entire time. The OME Modified scoring system includes variable ranges depending on the domain assessed. For attitude and attention, scores range from 1 to 7, with higher scores indicating better outcomes. For activity, scores range from 0 to 3, where a score of 3 represents a greater time the participant was manifesting the activites.

CONTACTS AND LOCATIONS:
Locations (1):
- Ridgewood Health Campus, Lawrenceburg, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified IPD that underlies the results reported in the primary publication. This includes individual-level data on demographics, baseline characteristics, outcome measures, and adverse events. Personally identifiable information will be removed to protect participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Unending (Beginning after the publication of our study, with no end date).
Access Criteria: Future doctor of occupational therapy students at Northern Kentucky University who are interested in further developing research in this domain will be able to access IPD and supporting information. They can access all supporting information via our password-protected flash drive, where we are storing all of the data and study information.

REFERENCES:
- See also: St. Louis School of Medicine: Cognitive Stimulation Therapy (CST) and Individual Cognitive Stimulation Therapy (iCST) — https://www.slu.edu/medicine/internal-medicine/geriatric-medicine/aging-successfully/cognitive-stimulation-therapy.php

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT06978972/Prot_SAP_005.pdf
  • Informed Consent Form: Participants ICF (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT06978972/ICF_003.pdf
  • Informed Consent Form: Participants with POAs ICF (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT06978972/ICF_004.pdf